CLINICAL TRIAL: NCT00612521
Title: Prophylactic Intra-coronary Adenosine to Prevent Post Coronary Artery Stenting Myonecrosis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: At half the sample size, the results were negative with no benefit demonstrated with adenosine.
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2007446-01H
Record Dates: First submitted 2008-01-25; First posted 2008-02-11 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Artery Stenosis; Coronary Artery Disease
Keywords: Coronary artery disease; Coronary artery stenting; peri-procedural myonecrosis; Adenosine
MeSH Terms: conditions — Coronary Stenosis; Coronary Artery Disease | interventions — Adenosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Either Placebo or Adenosine mixed with normal saline at a concentration of 6 micrograms per milliliter.
  Interventions: Drug: Adenosine
- 2 (Other): Either Placebo or Adenosine mixed with normal saline at a concentration of 6 micrograms per milliliter.
  Interventions: Drug: Adenosine

INTERVENTIONS:
Drug: Adenosine — For lesions in the left coronary system the patient will receive either 120 micrograms of adenosine in 20 mls of normal saline or placebo prior to the wiring, pre-dilatation, stenting and post-dilatation of the target coronary stenosis. For lesions in the right coronary system the patient will receive either 60 micrograms of adenosine in 10 mls of normal saline or placebo prior to the wiring, pre-dilatation, stenting and post-dilatation of the target coronary stenosis.

SUMMARY:
Myocardial damage occurs in up to 40% of cases when sensitive biomarkers are measured after coronary artery stenting. Such events have been associated with poor outcomes both at 30 days and long term. The cause of such damage is multi-factorial and includes distal propagation of atheromatous and thrombotic debris and the subsequent infiltration of the microcirculation with inflammatory cells. Individually or together these events can occlude the micro-circulation and lead impaired blood flow to heart muscle.

The vasodilator adenosine is commonly used in cases of impaired flow in an endeavor to improve flow rate and limit myocardial damage. Unfortunately the efficacy of this therapy is limited. More recently, there have been clinical studies looking at the administration of adenosine before any potential damage by ballooning or stenting, in an effort to avoid poor distal flow post procedure and thus limit any myocardial damage. Although small numbers of subjects have been included in these trials, there have been encouraging preliminary data.

The aim of this study is to assess whether the use of intra-coronary adenosine given directly into the target coronary artery prior to stenting can reduce the incidence of myonecrosis (heart muscle damage)over placebo. We also aim to assess whether this translates to better outcomes at 30 day follow up.

DETAILED DESCRIPTION:
Prior clinical studies looking at the administration of adenosine before coronary artery stenting have looked at small numbers of subjects and did not mandate previous statin therapy or high dose loading of clopidogrel before stenting, both of which can also help lower the rate of peri-procedural myonecrosis.

Our aim is to assess the above mentioned therapy in patients on optimal treatment with statins, dual antiplatelet agents and standard of care anti-coagulants.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing percutaneous coronary balloon angioplasty and stenting
* Ages 18 years and older
* TIMI III flow on the initial angiography
* Native coronary artery lesions

Exclusion Criteria:

* Patients unable to give consent
* Adenosine allergy
* Severe asthma with bronchial reactivity
* Cardiogenic or circulatory shock
* Acute or chronic total coronary artery occlusions
* Patients requiring Rotablator therapy
* In stent restenosis
* Second or third degree AV block without a permanent pacemaker
* ST-Elevation MI
* Elevated baseline CK/ CK-MB or troponin levels (Pre-existing Non-STemi)
* Current pregnancy
* Patients not already on statin therapy or intolerant of statins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-08; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Peri-procedural myocardial infarction | 24 hours post procedure

SECONDARY OUTCOMES:
TIMI frame count | Final angiographic picture during the index procedure
Death, myocardial infarction or target lesion revascularization | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Marino Labinaz, MD FRCP, Principal Investigator — Director of Interventional Cardiology - University of Ottawa Heart Institute
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada